CLINICAL TRIAL: NCT02988349
Title: Ecological Effect of 8% Arginine Dentifrice on Oral Microbiota of Caries-Free and Caries-active Populations
Brief Title: Ecological Effect of Arginine Dentifrice on Oral Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Xin Xu, Clinical Professor, Sichuan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCHSIRB-D-2013-067-R2
Record Dates: First submitted 2016-11-24; First posted 2016-12-09 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-04

CONDITIONS: Dental Caries; Oral Bacterial Infection; Microbiota
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caries-free subjects (Active Comparator): Subjects will use Colgate® Sensitive Pro-Relief® toothpaste for 2 weeks,.
  Interventions: Other: Colgate® Sensitive Pro-Relief® toothpaste
- Caries-active subjects (Experimental): Subjects will use Colgate® Sensitive Pro-Relief® toothpaste for 2 weeks,.
  Interventions: Other: Colgate® Sensitive Pro-Relief® toothpaste

INTERVENTIONS:
Other: Colgate® Sensitive Pro-Relief® toothpaste — Subjects will be instructed to brush their teeth twice daily for 3 min using Colgate® Sensitive Pro-Relief® toothpaste for 2 weeks.

SUMMARY:
caries-free (CF) individuals caries-active (CA) individuals (DMFT ≥ 6) will be recruited. Subjects will be instructed to brush their teeth twice daily for 3 min using Colgate® Sensitive Pro-Relief® toothpaste (containing 8% arginine and 1450 ppm NaF) for 2 weeks. Supra- and subgingival plaque, saliva, and in situ plaque samples will be collected before and after the treatment for laboratory analyses.

DETAILED DESCRIPTION:
21 caries-free (CF) individuals with no clinical evidence of caries experience [decayed, missing and filled teeth (DMFT) = 0] and 21 caries-active (CA) individuals (DMFT ≥ 6) will be recruited in the clinical trial. The exclusion criteria are: smoker or former smoker, presence of any systemic disease that could alter the production or composition of saliva, treatment with antibiotics, steroids or any medication known to cause dry mouth in the last 3 months, and presence of dental prostheses or orthodontic devices. Subjects will be instructed to brush their teeth twice daily for 3 min using Colgate® Sensitive Pro-Relief® toothpaste (containing 8% arginine and 1450 ppm NaF) for 2 weeks. Volunteers are asked to refrain from brushing and flossing their teeth, eating, and drinking anything other than water for 12 h prior to sample collection visits at the end of both phases. Supra- and subgingival plaque (15 subjects in each group), saliva (21 subjects in each group), and in situ plaque samples (3 subjects in each group) will be collected before and after the treatment. Scraped plaque and saliva samples will be immediately transferred to and dispersed in sterile micro-centrifuge tubes containing 1×phosphate-buffered saline (PBS), and stored at -80 °C until needed for analysis. The in situ plaque samples will be transferred into 4% paraformaldehyde, kept under 4 °C for 16 h, and then stored in 50% (v/v) ethanol at -20 °C.

ELIGIBILITY:
Inclusion Criteria:

* caries-free individuals with no clinical evidence of caries experience [decayed, missing and filled teeth (DMFT) = 0] and caries-active individuals (DMFT ≥ 6) were recruited

Exclusion Criteria:

* smoker or former smoker, presence of any systemic disease that could alter the production or composition of saliva, treatment with antibiotics, steroids or any medication known to cause dry mouth in the last 3 months, and presence of dental prostheses or orthodontic devices.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xin Xu, D.D.S, Principal Investigator — West China Hospital of Stomatology, Sichuan University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first recruitment took place on Oct. 2013, in the Department of Operative Dentistry and Endodontics, West China Hospital of Stomatology. 15 CF and 15 CA individuals were recruited by the end of Nov. 2013.
  The second recruitment took place on May in the same location. 2014. 6 CF and 6 CA individuals were recruited by the end of Jun. 2014.
Period: Overall Study
Arm/Group | Caries-free Subjects | Caries-active Subjects
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caries-free Subjects | Caries-active Subjects | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 23 [19 to 31] | 23 [19 to 28] | 23 [19 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 17 | 28
  Male | 10 | 4 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  China | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: The Change of Abundance of Specific Oral Microbes After Intervention as Assessed by 16S rRNA Sequencing
Description: Saliva and dental plaque samples will be collected, and the abundance of specific oral microbes such as Streptococcus mutans, Streptococcus sanguinis will be quantified by microbial 16S rRNA sequencing.
Time Frame: baseline , 2 week
Measure: Mean (Standard Deviation); unit: percentage of bacteria
Arm/Group | Caries-free Subjects | Caries-active Subjects
Number analyzed (Participants) | 21 | 21
percentage of bacteria
  Baseline: sm in supragingival plaque | 0.00756 (0.00726) | 0.14636 (0.23221)
  Baseline: sm in subgingival plaque | 0.00629 (0.00835) | 0.11956 (0.20686)
  Baseline: sm in saliva | 0.00608 (0.00575) | 0.01314 (0.01272)
  Baseline: ss in supragingival plaque | 1.007766667 (1.168793223) | 0.521506667 (0.511640082)
  Baseline: ss in subgingival plaque | 2.064646667 (2.595662011) | 1.539913333 (1.369851357)
  Baseline: ss in saliva | 0.812706667 (1.040344461) | 0.18324 (0.199811864)
  2 week: sm in supragingival plaque | 0.003406667 (0.003320384) | 0.009526667 (0.011458775)
  2 week: sm in subgingival plaque | 0.0033 (0.006143173) | 0.00284 (0.005101792)
  2 week: sm in saliva | 0.002493333 (0.004110347) | 0.003006667 (0.002304488)
  2 week: ss in supragingival plaque | 1.655106667 (1.274066247) | 3.21486 (3.436273455)
  2 week: ss in subgingival plaque | 4.588546667 (4.92217214) | 3.232233333 (3.336652867)
  2 week: ss in saliva | 1.3109 (0.885269549) | 2.040286667 (3.369773515)

2. Secondary Outcome: The Change of Relative Activities of Microbial Enzymes After Intervention as Determined by Laboratory Enzymatic Assays
Description: Saliva and dental plaque samples will be collected and microbial enzyme activity will be quantified in the lab. Measures include relative enzyme activity of arginine deiminase, urease and lactase dehydrogenase as determined by standard laboratory enzymatic assay protocols.
Time Frame: baseline ,2 week
Population: Among the 21 participants in each group，we only measured the enzyme activity from randomly choosed 15 participants from each group.
Measure: Mean (Standard Deviation); unit: enzyme activity (μmol/min/g)
Arm/Group | Caries-free Subjects | Caries-active Subjects
Number analyzed (Participants) | 15 | 15
enzyme activity (μmol/min/g)
  baseline: ADS activity in supragingival plaque | 0.8945 (0.13310) | 0.3653 (0.06108)
  baseline: ADS activity in subgingival plaque | 0.63150 (0.08604) | 0.29110 (0.04347)
  baseline: ADS activity in saliva plaque | 0.75870 (0.09211) | 0.23470 (0.03328)
  baseline: urease activity in supragingival plaque | 0.6795 (0.11518) | 0.3207 (0.06317)
  baseline: urease activity in subgingival plaque | 0.71840 (0.08770) | 0.34630 (0.04611)
  baseline: urease activity in saliva | 0.72900 (0.66210) | 0.17920 (0.03047)
  baseline: LDH activity in supragingival plaque | 8.859050 (0.6648584) | 20.965090 (1.549900)
  baseline: LDH activity in subgingival plaque | 7.267220 (0.2555969) | 17.576110 (0.887500)
  baseline: LDH activity in saliva | 7.508787 (0.8707994) | 16.053870 (2.361490)
  2 week: ADS activity in supragingival plaque | 1.0771 (0.23754) | 0.8418 (0.13711)
  2 week: ADS activity in subgingival plaque | 0.74650 (0.10275) | 0.73600 (0.07218)
  2 week: ADS activity in saliva | 0.77410 (0.11136) | 0.34850 (0.04391)
  2 week: urease activity in supragingival plaque | 0.5871 (0.07970) | 0.6508 (0.10083)
  2 week: urease activity in subgingival plaque | 0.73330 (0.06165) | 0.69680 (0.08427)
  2 week: urease activity in saliva | 0.73240 (0.05464) | 0.25260 (0.04560)
  2 week: LDH activity in supragingival plaque | 11.347060 (0.9240766) | 14.096910 (0.3565668)
  2 week: LDH activity in subgingival plaque | 8.664124 (0.8184378) | 11.649030 (1.135210)
  2 week: LDH activity in saliva | 9.496731 (0.1797688) | 15.268450 (0.3687766)

ADVERSE EVENTS:
Arm/Group | Caries-free Subjects | Caries-active Subjects
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No